CLINICAL TRIAL: NCT05286658
Title: Behavioral and Neural Measures of Speech Motor Control
Brief Title: Behavioral and Neural Responses to External Alterations of Speech Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-1128 MEG Imaging (Exp 5); Protocol Version 8/25/2021 (Other: UW Madison); A481800 (Other: UW Madison); 1R01DC019134-01A1 (NIH)
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Speech
Keywords: speech motor control; vocal learning
MeSH Terms: conditions — Speech | interventions — Magnetoencephalography; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Adult Speakers (Experimental): healthy adult participants across the lifespan in three groups:18-35, 36-55, and 56+
  Interventions: Behavioral: MEG/EEG; Behavioral: MRI; Behavioral: Speaking Tasks

INTERVENTIONS:
Behavioral: MEG/EEG — The participant will sit still while their head is slid into the helmet-shaped bottom of the MEG device. The MEG contains sensors that passively detect weak magnetic fields outside the head produced by brain activity. The computer records the brain's electrical activity on the screen as wavy lines. The investigators will also ask you to wear sensors to capture eye-blinks (electrooculogram) and heartbeats (electrocardiogram) to facilitate removal from the MEG signal during analysis.
  Participant will sit in front of a projector screen and be asked to put on a pair of headphones. Participant will be shown real words or nonsense words to read, the investigators may play sounds through headphones for the participant to repeat. Participant speech will be recorded by a microphone. The investigators may ask the participant to identify what they heard by pressing a button on a button-box. These tasks are expected to take about one hour to complete.
  Other Names: magnetoencephalogram / electroencephalogram
Behavioral: MRI — An MRI is a test that uses a magnetic field and pulses of radio wave energy to make pictures of organs and structures inside the body. The participant will be able to hear and speak to the research staff at all times during the MRI procedures. The MRI test will take about 15 minutes.
  Other Names: magnetic resonance imaging
Behavioral: Speaking Tasks — The participant may be asked to perform some of the tasks from MEG again, this time outside of the scanner. As before, the participant may see real words or nonsense words to read, and the investigators may play sounds through headphones and ask the participant to repeat them. Participant speech will be recorded by a microphone. The investigators may ask the participant to identify what they heard by pressing a button on a button-box. These tasks are expected to take about one hour to complete.

SUMMARY:
The purpose of this research study is to understand how the brain processes and controls speech in healthy people. The investigators are doing this research because it will help identify the mechanisms that allow people to perceive their own speech errors and to learn new speech sounds, which may be applied to people who have communication disorders. 15 participants will be enrolled into this part of the study and can expect to be on study for 3-4 visits of 2-4 hours each.

DETAILED DESCRIPTION:
The overall study (Establishing the clinical utility of sensorimotor adaptation for speech rehabilitation) aims to understand how cognitive, perceptual, and motor processes are integrated in the control of speech movements. The investigators study how this complex skill is performed in healthy speakers to understand how this system functions, how this skill relates to the perception of speech, and what role different parts of the brain play in this process. Different studies look at how speech motor control is executed, maintained, and changed. Overall, the study will recruit 329 participants over the course of 5 years. Participants can expect to be on study for up to 3 weeks.

The entire study is composed of 8 experiments and 6 interventions. The present record represents the experiments involving magnetoencephalographic (MEG) imaging, i.e. Experiment 5: Behavioral and neural responses to external alterations of speech variability.

This paradigm modulates the perceived speech variability of participants through three different altered auditory feedback sessions: an inward-pushing feedback perturbation that decreases perceived variability by playing back participants' speech closer to the center of their vowel distributions, an outward-pushing feedback perturbation that increases perceived variability by playing back participants' speech farther from the center of their vowel distributions, and a normal feedback condition in which speech feedback is played back without perturbation. Participants will complete this paradigm during MEG imaging, which will noninvasively measure auditory cortical activity evoked during speech production and playback.

ELIGIBILITY:
Inclusion Criteria (Patients):

* English-speaking adults
* diagnosed communicative disorder, target populations may include:

  * stroke survivors with aphasia
  * individuals with cerebellar ataxia
  * individuals with parkinson's disease
  * individuals who use cochlear implants to hear
  * adults who stutter

Inclusion Criteria (Control):

* English-speaking adults
* normal hearing and speech
* no history of stroke or neurological conditions

Exclusion Criteria:

* Native language other than English
* Any neurological disorders other than the disorder of interest
* Any history of hearing disorders
* Uncorrected vision problems that prevent participants from seeing visually-presented stimuli
* Significant cognitive impairments that prevent participants from carrying out the task or from giving informed consent
* Vulnerable populations (minors and prisoners)
* Additional exclusionary criteria if participating in neuroimaging:

  * Implanted paramagnetic materials (metal clips, plates, pacemakers, etc.)
  * Head too large for MEG recording helmet
  * Claustrophobia or intolerance of MRI scanner noise
  * Low signal to noise ratio in pilot MEG recordings
  * High levels of artifacts (eye-blinks, etc.)
  * Inability to produce the speech sounds proposed with minimal movement
  * Left-handedness
* Additional exclusionary criteria if participating in transcranial magnetic stimulation (TMS):

  * Implanted paramagnetic materials (metal clips, plates, pacemakers, etc.)
  * Increased risk in the event of a seizure
  * Serious heart disease
  * Increased intracranial pressure
  * Pregnancy
  * History of seizures
  * Family history of epilepsy
  * Epileptogenic medications
  * Chronic or transient disruption of sleep (including jet lag)
  * History of fainting
  * Chronic or transient increase in stressful experiences
  * Use of illegal drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Niziolek, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Link to study record for experiment 7 [NCT05723575] — https://clinicaltrials.gov/study/NCT05723575

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adult Speakers: Healthy adult participants across the lifespan.
  The participant will sit still while their head is slid into the helmet-shaped bottom of the MEG device. The MEG contains sensors that passively detect weak magnetic fields outside the head produced by brain activity. The computer records the brain's electrical activity on the screen as wavy lines.
  Participant will sit in front of a projector screen and be asked to put on a pair of headphones and be asked to read words or repeat sounds into a microphone. These tasks are expected to take about one hour to complete.
  The participant will undergo MRI scans and be able to hear and speak to the research staff at all times during the MRI procedures. The MRI test will take about 15 minutes.
  Speaking Tasks: The participant may be asked to perform some of the tasks from MEG again, this time outside of the scanner. These tasks are expected to take about one hour to complete.
Period: Overall Study
Arm/Group | Healthy Adult Speakers
Started | 17
Inward Variability Condition | 15
Outward Variability Condition | 15
Control Condition | 15
Analysis Population | 15
Completed | 15
Not Completed | 2
Not completed — Head circumference too large for MEG scanner (exclusion criterion for the study). | 1
Not completed — Participant did not show SIS (the dependent measure), thus the hypothesis could not be assessed | 1

BASELINE CHARACTERISTICS:
Population: Participants with measurable neural suppression (relevant outcome measure)
Groups:
- Healthy Adult Speakers: Healthy adult participants across the lifespan.
  Interventions: This paradigm modulates the perceived speech variability of participants through three different altered auditory feedback sessions: an inward-pushing feedback perturbation that decreases perceived variability by playing back participants' speech closer to the center of their vowel distributions, an outward-pushing feedback perturbation that increases perceived variability by playing back participants' speech farther from the center of their vowel distributions, and a normal feedback condition in which speech feedback is played back without perturbation. The participants completed all three sessions during magnetoencephalographic (MEG) imaging, which noninvasively measured auditory cortical activity evoked during speech production and playback.
Arm/Group | Healthy Adult Speakers
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Speaking-Induced Suppression (SIS) Change, Defined as the Percent Change of SIS (the Z-score Difference in Average M100 Amplitude in the Speak Condition Compared With the Listen Condition) From Baseline to Test Phases
Description: The dependent measure is the speaking-induced suppression (SIS) defined as the z-score difference in average M100 amplitude in the speak condition compared with the listen condition. The M100 peak is defined as the peak activity between 75 and 150 ms after stimulus onset; peaks will be confirmed by visual inspection. The percent change in this SIS from the pre-test (baseline phase at the beginning of the MEG scan) to the post-test (test phase at the end of the MEG scan) is evaluated for each of three visits: "in", "out", and "control".
Time Frame: Data were collected over 3 individual hour-long MEG sessions over 3 weeks (pre-test vs. post-test compared within the same session).
Measure: Mean (Standard Deviation); unit: percent change (of z-score difference)
Arm/Group | Healthy Adult Speakers
Number analyzed (Participants) | 15
percent change (of z-score difference)
  "In": inward variability condition | 7.4 (16.1)
  "Out": outward variability condition | -22.2 (8.2)
  "Control": control condition | 28.9 (15.6)

ADVERSE EVENTS:
Time Frame: Subjects participated in four sessions (3 1-hour MEG scans and 1 1-hour behavioral visit) over the course of one month.
Description: Minimal risk basic science study, no adverse event collection plan required
Groups:
- Healthy Adult Speakers: Healthy adult participants across the lifespan.
Arm/Group | Healthy Adult Speakers
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT05286658/Prot_SAP_000.pdf